CLINICAL TRIAL: NCT03159377
Title: Ultra-Low Dose CT Denoising for Lung Nodule Detection
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Edith Marom, Professor, Sheba Medical Center
Other Study IDs: SHEBA - 16- 3651- EM - CTIL
Record Dates: First submitted 2017-05-17; First posted 2017-05-18 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Nodule, Multiple
Keywords: pulmonary nodule, CT, low dose
MeSH Terms: conditions — Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients scheduled for a chest CT: Inpatients or outpatients scheduled for a chest CT in our medical center
  Interventions: Device: Ultra low dose chest CT

INTERVENTIONS:
Device: Ultra low dose chest CT — Performing an ultra low dose chest CT (ULDCT) in addition to a clinically indicated chest CT and assessing nodule detection with a recently developed denoising algorithm

SUMMARY:
We will perform an ultra low-dose CT (ULDCT) in addition to a regular chest CT scan for adult patients undergoing a clinically indicated chest CT. Using a recently developed computationally efficient algorithm for the denoising of ULDCT scans after image reconstruction, we will compare the sensitivity, specificity and accuracy of lesion detection with the ULDCT as compared to the regular CT scan.

DETAILED DESCRIPTION:
Patient cohort: Two hundred patients will be recruited for this study. Patients will be comprised of two groups: an inpatient group of patients from the Internal Medicine Department E for which a chest CT is ordered during their hospitalization; and ambulatory patients arriving for an ambulatory chest CT in the early afternoon. The treating clinician ordering the chest CT for the patients from Internal Medicine E will consent the inpatients while a chest radiologist from the Radiology Department will consent the outpatients arriving in the early afternoon for a chest CT study. For inclusion in the study, patients will be adults, older than 18 years old with the ability to follow orders and hold their breath for 8 seconds as determined by the physician at time of study consent.

Imaging method: All patients consented for this study will be imaged on a dedicated scanner for the study, Revolution (GE, Milwaukee, WI). Immediately following the patient's diagnostic chest CT scan, an ultra low dose chest CT scan will be obtained. The routine CT scans of the patients consented for this study will be performed using our routine protocol on the GE Revolution which typically delivers at our institution an average effective dose of 2.9mSv (range 0.95-3.01mSv) while our other Philips routine chest CT scan delivers an average effective dose of 10.5mSv (range 10.29-12.95mSv). With the addition of the ultra low dose technique, which delivers a radiation dose of a range of 0.5-1 mSv (calculated from a pilot study we obtained on pigs), patients are expected to get an total radiation dose for both scans together of about 4 mSv which is less than 10.5mSv (the normal dose for the Phillips CT machine at our institution). Just as a comparison, a meticulous study looking at multiple institutions showed that the average effective dose from a routine chest CT is 7mSv, range 4-18mSv and for a chest CT with pulmonary embolism protocol an average effective dose of 15mSv with a range of 13-40mSv .

Image evaluation: The diagnostic chest CT scan will be sent to the PACS as usual and interpreted immediately, during the same day, as per normal inpatient clinical operations protocol at our institution. The ultra low dose CT scan will be automatically sent to the computational imaging lab processing station, which will denoise the image. After denoising the images will be automatically forwarded to the PACS under the same accession number of the routine chest CT scan. Comparison of the ultra low dose denoised images to the routine chest CT images will be performed by an experienced chest radiologist at a later date, at least one week after date of acquisition to prevent any memorability of the original image. Radiologists' memory of findings has been shown to be poor, even when viewed immediately but slightly worse when time passes [Evans]. The radiologist will document the presence of nodules, consolidation, ground glass opacities, emphysema, fibrosis with abnormalities marked on the images in the PACS. Following completion of the table, the routine chest CT scan will be used as the gold standard for the presence of the imaging findings. The documented ultra low dose CT findings will be compared to the images from the routine chest CT scans. Each finding documented will be individually documented as a true finding if also seen on the routine chest CT scan or false finding if not present on the routine chest CT scan. Additional findings only seen on the routine chest CT scan will be documented as missed findings.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient scheduled for a chest CT, in-patient or outpatient

Exclusion Criteria:

* Children

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any adult patient scheduled for a chest CT, in-patient or outpatient, in our institution
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Identification of a pulmonary nodule | Patient collection in two years
  Comparison of sensitivity, specificity and accuracy in identifying a pulmonary nodule when comparing denoised ULDCT to a regular CT.

CONTACTS AND LOCATIONS:
Overall Officials: Edith M Marom, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided
The only specific data of this study is low dose CT images while everything else is patient's usual care and not part of the study. Have not decided who may or may not use our low dose images.